CLINICAL TRIAL: NCT07170228
Title: The Effects of Casein Supplementation Timing on Exercise Performance: A Comparison Between Pre-Sleep and Post-Exercise Intake
Brief Title: Casein Supplementation: Pre-Sleep vs. Post-Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Serdar Bayrakdaroğlu (Other)
Responsible Party: Sponsor-Investigator, Serdar Bayrakdaroğlu, Associate Professor, Principal Investigato, Gümüşhane Universıty
Organization: Gümüşhane Universıty (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: GTU-2025-CASEIN01; Ethics Committee -GTU-EC-2024 (Other: Gumushane University)
Record Dates: First submitted 2025-09-05; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Athletic Performance
Keywords: Casein Supplementation; Pre-Sleep Protein Intake; Post-Exercise Protein Intake; Muscle Recovery; Anaerobic Performance

STUDY DESIGN:
Intervention Model Description: Participants were randomized into three parallel groups: pre-sleep casein ingestion, post-exercise casein ingestion, or control, using stratified block randomization.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors were blinded to participant group assignments, while participants and investigators were not blinded due to the nature of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pre-Sleep Casein Ingestion Group (Experimental): Participants consumed 30 g of micellar casein dissolved in 300 mL of water 30-60 minutes before sleep following the standardized high-intensity resistance training session. Supplement intake was directly monitored by the research team to ensure compliance.
  Interventions: Dietary Supplement: Micellar Casein
- Post-Exercise Casein Ingestion Group (Experimental): Participants consumed 30 g of micellar casein dissolved in 300 mL of water 10-15 minutes after completing the standardized high-intensity resistance training session. Supplement preparation and intake were supervised by the research team.
  Interventions: Dietary Supplement: Micellar Casein
- Control Group (No Intervention): Participants completed the standardized high-intensity resistance training protocol but did not receive any supplementation.

INTERVENTIONS:
Dietary Supplement: Micellar Casein — Participants consumed 30 g of micellar casein powder dissolved in 300 mL of water.
  Supplement timing varied by group:
  Post-Exercise Casein Ingestion Group (PECIG): Taken 10-15 minutes after completing the standardized high-intensity resistance training session.
  Pre-Sleep Casein Ingestion Group (PSCIG): Taken 30-60 minutes before bedtime on the same day as the training session.
  The control group received no supplementation. All supplements were prepared and monitored by the research team to ensure dosage accuracy and participant compliance.
  Arms: Post-Exercise Casein Ingestion Group; Pre-Sleep Casein Ingestion Group

SUMMARY:
This randomized controlled trial aimed to investigate the effects of casein supplementation timing on post-exercise recovery and exercise performance in trained football players. Participants were allocated into three groups: pre-sleep casein ingestion, post-exercise casein ingestion, and control. The study compared the effects of pre-sleep and post-exercise casein intake on anaerobic performance, agility, and recovery markers following a standardized high-intensity resistance training session.

DETAILED DESCRIPTION:
Casein is a slow-digesting protein commonly used as a dietary supplement to promote muscle recovery and adaptation. Although casein is traditionally consumed before sleep to maximize overnight muscle protein synthesis, limited evidence exists regarding the optimal timing of casein ingestion relative to exercise.

This study employed a randomized controlled experimental design to compare the effects of pre-sleep versus post-exercise casein supplementation on recovery and performance outcomes in trained football players. Twenty-four male participants were stratified by playing position (defender, midfielder, forward) and randomized into three groups: pre-sleep casein ingestion group (PSCIG), post-exercise casein ingestion group (PECIG), and control group (CG). All participants first completed a familiarization session and pre-test assessments, including the countermovement jump (CMJ), Illinois Agility Test, and Running-based Anaerobic Sprint Test (RAST).

After the pre-tests, all players performed a standardized high-intensity resistance training protocol designed to induce muscle fatigue. Participants in the PECIG consumed 30 g of micellar casein dissolved in 300 mL of water within 10-15 minutes post-exercise, while participants in the PSCIG consumed the same supplement 30-60 minutes before sleep. The control group did not receive any supplementation. Twenty-four ± 1 hours after the resistance training, post-tests were conducted using the same protocols as the pre-tests.

The primary aim of this study was to determine whether casein supplementation timing (pre-sleep vs. post-exercise) differentially influences recovery and subsequent anaerobic performance. Outcomes from this trial may provide practical recommendations for athletes and coaches regarding optimal protein supplementation strategies to enhance recovery and performance.

ELIGIBILITY:
Inclusion Criteria:

* Male football players aged 18 to 25 years.
* At least three years of competitive soccer experience.
* Engaged in structured soccer training at least three times per week during the previous six months.
* Clearance to participate based on the Physical Activity Readiness Questionnaire (PAR-Q) (Thomas et al., 1992; Bredin et al., 2013).
* Provided written informed consent prior to participation.

Exclusion Criteria:

* Any musculoskeletal injury or surgery within the past six months.
* Reported milk or casein intolerance or allergy.
* Regular use of ergogenic supplements such as protein or creatine during the previous four weeks
* Medical conditions or limitations that could interfere with maximal exercise performance.
* Non-compliance with study procedures or training/testing protocols.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-03-14 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
Peak Power (RAST Test) | Change from baseline (pre-test) to 24 hours post-training (post-test)
  Peak power will be calculated using body mass and sprint times obtained during the RAST test to assess maximal anaerobic performance. Measurements will be taken at baseline and 24 hours post-training.

SECONDARY OUTCOMES:
Mean Power (RAST Test) | Change from baseline (pre-test) to 24 hours post-training (post-test)
  Mean power will be calculated from total sprint time and body mass during the Running-based Anaerobic Sprint Test (RAST) to evaluate anaerobic endurance performance. Measurements will be collected pre- and 24 hours post-training.
Fatigue Index (RAST Test) | Change from baseline (pre-test) to 24 hours post-training (post-test)
  Fatigue index will be calculated using the difference between the highest and lowest sprint times divided by the total sprint time during the RAST test. It reflects fatigue and recovery capacity. Measurements will be collected pre- and 24 hours post-training.
Countermovement Jump (CMJ) Height | Change from baseline (pre-test) to 24 hours post-training (post-test)
  CMJ height will be measured using a validated jump mat system to assess lower-limb explosive power. Measurements will be collected pre- and 24 hours post-training under standardized conditions.
Illinois Agility Test Time | Change from baseline (pre-test) to 24 hours post-training (post-test)
  Agility performance will be assessed using the Illinois Agility Test to evaluate change of direction speed and overall agility. Measurements will be collected pre- and 24 hours post-training under standardized environmental conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- Gumushane University, Faculty of Sport Sciences, Gümüşhane, Gümüşhane Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because of privacy concerns and restrictions imposed by the ethics committee approval.